CLINICAL TRIAL: NCT02545998
Title: Conducting Annual Asthma Reviews Using Telehealthcare: Comparison With Standard Care (Face-to-face Consultations)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15IC2535
Record Dates: First submitted 2015-05-21; First posted 2015-09-10 (Estimated); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Asthma
Keywords: Telehealthcare
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): Patients will receive a face-to-face asthma review
- Telehealthcare (Active Comparator): Patients will receive a telephone consultation and e-mail with attached PAAP and video link
  Interventions: Other: Telehealthcare

INTERVENTIONS:
Other: Telehealthcare — Telephone consultation plus e-mail with attached PAAP and video link
  Arms: Telehealthcare

SUMMARY:
The National Report of Asthma Deaths published in 2014 highlighted significant deficiencies in both primary and secondary care resulting in one of the highest mortality rates in Europe. A key recommendation in the report is the provision of an annual asthma review in primary care.

Telehealthcare is an alternative means of service delivery incorporating the use of telephone and e-mail consultations which may improve access and quality of patient care. There is scant data on the role of teleheathcare in asthma care.

This is a single-centre, primary care-based, randomized controlled trial to evaluate the use of telehealthcare to conduct the annual asthma review for adult patients with well-controlled asthma. This will be compared with standard care (face-to-face consultations).

Telehealthcare will consist of a telephone consultation followed by an e-mail with an attached personalised asthma action plan and a link to a video demonstrating inhaler technique.

Standard care will involve a face-to-face consultation in primary care. The two patient groups will be compared prospectively to determine whether there is a difference in the quality of care evaluated in terms of the patient experience/ satisfaction, health-related quality of life, asthma control and frequency of asthma exacerbations over a 6 month period after the asthma review.

The data will be presented in the form of frequency tables, bar charts and pie charts. Non-parametric tests will be applied to determine whether there is a significant difference in the quality of care received.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over, registered at Balham Park Surgery
* Patients diagnosed with asthma (patients on the asthma register)
* Patients with well-controlled asthma (ACT score 20 and over; no out of hours/ A&E attendances/ PO steroids/ hospital admissions since the last asthma review in primary care)

Exclusion Criteria:

* Patients aged less than 18
* Patients with poorly controlled asthma (ACT score 19 or less; out of hours/ A&E attendance/ hospital admission/ PO steroids since last asthma review in primary care)
* Patients with a mental health diagnosis
* Patients without an up to date contact telephone number or with communication difficulties that would prevent or restrict their use of the technology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Glynne, MRCP MRCGP, Principal Investigator — Balham Park Surgery, Wandsworth CCG
Locations (1):
- Balham Park Surgery, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care: Patients received a face-to-face asthma review
- Telehealthcare: Patients received a telehealthcare asthma review consisting of a telephone consultation and an e-mail with attached PAAP and video link.
Period: Overall Study
Arm/Group | Standard Care | Telehealthcare
Started | 44 | 44
Received the Intervention | 33 | 42
Completed | 29 | 39
Not Completed | 15 | 5
Not completed — Lost to Follow-up | 12 | 3
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Telehealthcare | Total
Number analyzed (Participants) | 33 | 42 | 75
Age, Customized [Median (Inter-Quartile Range); unit: years] | 38.0 [30.0 to 48.0] | 38.5 [30.0 to 50.0] | 38.0 [30.0 to 50.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 44
  Male | 13 | 18 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  White | 29 | 40 | 69
  Non-white | 4 | 2 | 6
Occupation [Number; unit: participants]
  Employed/ full time education | 29 | 37 | 66
  Unemployed/ retired | 4 | 5 | 9
Median ACT score [Median (Inter-Quartile Range); unit: units on a scale] — Asthma Control Test (ACT) was used to screen patients for poor asthma control prior to study enrolment. This is a simple, five-item, validated questionnaire that is designed to identify patients (>12 years old) with poorly controlled asthma. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
  units on a scale | 24 [22 to 25] | 23 [21 to 25] | 23 [22 to 25]
Median AQLQ score [Median (Inter-Quartile Range); unit: units on a scale] — Asthma Quality of Life Questionnaire (AQLQ) is a valid, reliable questionnaire that measures the "functional problems" (physical, emotional, social and occupational) that are most troublesome to adults aged 17-70 years with asthma. For the purpose of this study, a 15-item mini-AQLQ was used, with scores ranging from 1 (severely impaired) to 7 (not impaired at all).
  units on a scale | 5.9 [5.4 to 6.6] | 6.2 [5.8 to 6.7] | 6.2 [5.53 to 6.6]
Median length of time since last asthma review [Median (Inter-Quartile Range); unit: months] | 32 [13 to 60] | 25 [17 to 60] | 30 [13 to 60]

OUTCOME MEASURES:

1. Primary Outcome: Patient Experience: Overall Patient Experience Score (General Practice Assessment Questionnaire GPAQ Score)
Description: General Practice Assessment Questionnaire (GPAQ) is a widely used questionnaire to assess the patient experience of general practice in the UK. It is designed to measure satisfaction across four domains: communication (8 items), confidence (3 items), access to care (2 items) and overall satisfaction (2 items). Patients rate their experience by selecting not of usually 5 responses (1= very good to 5= very poor). Response items were linearly rescaled to a 0-100 range (100 = most favourable response). 'Does not apply' responses were excluded from the analysis.
  This yielded four median domain scores for each patient (range 0-100 per domain).
  An overall patient experience score was calculated for each patient by adding the four domain scores together to give a total score out of 400 (range 0-400).
  The median overall patient experience score (+/- interquartile range) was calculated for each group and the scores were compared (tele healthcare vs control)
Time Frame: Up to 2 weeks after the asthma review
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Care | Telehealthcare
Number analyzed (Participants) | 33 | 42
score on a scale | 390.0 [367.5 to 400.0] | 400.0 [377.5 to 400.0]
Statistical Analysis 1: Comparison: Standard Care vs Telehealthcare; Test type: Superiority; p = 0.510, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Dropout Rate
Description: The dropout rate is the number of patients that failed to attend for an asthma review ('Did not attend', lost to follow up, or withdrew consent) in each patient group.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Telehealthcare
Number analyzed (Participants) | 44 | 44
Participants | 11 | 2
Statistical Analysis 1: Comparison: Standard Care vs Telehealthcare; Test type: Superiority; p = 0.014, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Average Consultation Length (Time)
Description: The average time taken for a standard asthma review vs a telehealthcare review will be recorded at the time of the asthma review
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Standard Care | Telehealthcare
Number analyzed (Participants) | 33 | 42
minutes | 20.0 [18.0 to 23.0] | 15.0 [12.0 to 17.0]
Statistical Analysis 1: Comparison: Standard Care vs Telehealthcare; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Health Related Quality of Life Score (Asthma Quality of Life Questionnaire (AQLQ))
Description: Quality of life will be assessed using the Asthma Quality of Life Questionnaire (AQLQ) in each group at the start of the study (before the asthma review) and 6 months after the asthma review.
  Asthma Quality of Life Questionnaire (AQLQ) is a valid, reliable questionnaire that measures the "functional problems" (physical, emotional, social and occupational) that are most troublesome to adults aged 17-70 years with asthma. For the purpose of this study, a 15-item mini-AQLQ was used, with scores ranging from 1 (severely impaired) to 7 (not impaired at all).
  The 6 month AQLQ score is presented in each group. The p value compares the change in AQLQ score from baseline to 6 months between the two groups.
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Care | Telehealthcare
Number analyzed (Participants) | 29 | 39
units on a scale | 6.4 [6.0 to 6.8] | 6.4 [6.1 to 6.8]
Statistical Analysis 1: Comparison: Standard Care vs Telehealthcare; Test type: Superiority; p = 0.589, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Asthma Control Test Score
Description: Assessment of asthma control using validated questionnaire at baseline (before the asthma review) and 6 months after the asthma review.
  The ACT score at 6 months is presented. The p value compares the change in ACT score from baseline to 6 months, in each group.
  Asthma Control Test (ACT) is a simple, five-item, validated questionnaire that is designed to identify patients (>12 years old) with poorly controlled asthma. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Time Frame: 6 months after asthma review.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Care | Telehealthcare
Number analyzed (Participants) | 29 | 39
score on a scale | 24 [23 to 25] | 23 [22 to 25]
Statistical Analysis 1: Comparison: Standard Care vs Telehealthcare; Test type: Superiority; p = 0.471, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Exacerbations.
Description: Number of exacerbations (unscheduled asthma consultations in primary care, courses of systemic steroids, out of hour attendances, hospital admissions) in the six months after the asthma review in each group.
Time Frame: In the six months after the asthma review.
Measure: Median (Inter-Quartile Range); unit: exacerbations
Arm/Group | Standard Care | Telehealthcare
Number analyzed (Participants) | 33 | 42
exacerbations | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Standard Care vs Telehealthcare; Test type: Superiority; p = 0.264, Sign test

7. Secondary Outcome: Future Preference
Description: After the asthma review, patients were asked whether they would prefer a tele healthcare asthma review in future.
  Percentage of patients that expressed preference for THC review is presented.
Time Frame: Within 2 weeks of the asthma review.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Telehealthcare
Number analyzed (Participants) | 33 | 42
Participants | 26 | 38

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Standard Care | Telehealthcare
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/42
Other Adverse Events (participants affected / at risk) | 0/33 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No